CLINICAL TRIAL: NCT05798442
Title: The Impact of Using a Smartphone Health Application in the Improvement of Cardiovascular Disease Risk Factors in the Omani Population; Prospective Randomized Clinical Trial
Brief Title: The Impact of Using a Smartphone Health Application in the Improvement of Cardiovascular Disease Risk Factors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Collaborators: Ministry of Higher Education, Research and Innovation (Ambiguous)
Responsible Party: Principal Investigator, Dr. Amani Alkhaifi, Principal Investigator, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Opulse app
Record Dates: First submitted 2023-03-12; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Hypercholesterolemia; Obesity; Diabetes Mellitus; Hypertension
Keywords: Mobile health application; Cardiovascular disease prevention; Metabolic risk factors; Behavioral risk factors
MeSH Terms: conditions — Hypercholesterolemia; Obesity; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Intervention Model Description: Patients with cardiovascular disease risk factors will be blindly randomized into two groups in a ratio of (1:1); mHealth app-based intervention group and a traditional mainstream face-to-face consultation group. The app-based intervention group will be given access to a mHealth app that will be specifically designed to motivate the users to increase their physical activity and healthy diet intake while reducing smoking and alcohol intake. The app provides the patients with standardized dietary and exercise guidelines and sends them frequent advice and reminders to follow the guidelines. Changes in the CVD risk factors of the participants will be assessed based on blood biochemical and anthropometric measurements collected every 4 months over a period of 20 months. The app will be designed to include interactive functions which allow the patients to insert their daily caloric intake and exercise, biometric data, track the improvement in their CVD risk factors and CVD risk score.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth app-based intervention group (Experimental): The app-based intervention group will be given access to a mHealth app that will be specifically designed to motivate the users to increase their physical activity and healthy diet intake while reducing smoking and alcohol intake. The app provides the patients with standardized dietary and exercise guidelines and sends them frequent advice and reminders to follow the guidelines. Changes in the CVD risk factors of the participants will be assessed based on blood biochemical and anthropometric measurements collected every 4 months over a period of 20 months. The app will be designed to include interactive functions which allow the patients to insert their daily caloric intake and exercise, biometric data, track the improvement in their CVD risk factors and CVD risk score.
  Interventions: Other: smartphone health application (Opulse)
- face-to-face consultation group (No Intervention): This group of patients will not have access to mHealth app and will receive the traditional face to face intervention.

INTERVENTIONS:
Other: smartphone health application (Opulse) — The Opulse app will be designed as a multifunction app that targets the modification of the behavioral and metabolic risk factors and provides comprehensive interventions for healthy diet, physical activity and smoking cessation among smokers.
  Arms: mHealth app-based intervention group

SUMMARY:
This study investigates the effectiveness of Mobile health application (mHealth apps) in the improvement of cardiovascular disease risk factors including metabolic and behavioral factors. The app will be tested on patients with any of the modifiable risk factors of CVD such as hypertension, obesity, hyperlipidemia, and impaired glycemic control/type 2 diabetes mellitus .

DETAILED DESCRIPTION:
The investigators aim in this study to reduce the risk of cardiovascular disease in patients with hypercholesterolemia, diabetes, obesity and hypertension. This will be achieved by motivating healthy lifestyle among the participants such as increasing physical activity and intake of healthy diet and reducing alcohol and tobacco consumption. The tool which will be used to motivate healthy lifestyle is a smartphone application which will be specifically designed to motivate behavioral change. Thus, the investigators hypothesis is that participants who have full access to the mobile application will show improved healthy lifestyle, reduced blood pressure, cholesterol and glucose and reduced BMI compared to the participants who don't have access to the mobile application.

ELIGIBILITY:
Inclusion Criteria:

* Presentation with at least one of the following metabolic abnormalities:
* Hypertensions (systolic blood pressure ≥ 130 mmHg and/or diastolic blood pressure ≥ 85 mmHg)
* Obesity (waist circumference ≥ 80 cm (women) or ≥ 94 cm (men) and BMI ≥ 25 kg/m2)
* Dyslipidemia (triglycerides ≥ 1.7 mmol/L or/and HDL-cholesterol ≤ 1.29 mmol/L (women) or ≤ 1.02 mmol/L (men) or/and LDL-Cholesterol > 5.18 mmol/L, serum total cholesterol ≥ 5.2 mmol/l)
* Impaired glycemia/type 2 diabetes (fasting plasma glucose ≥ 5.6 mmol/L)
* Arabic or English language speaking and able to read and write in one of these languages
* Possession of a smart mobile phone Willing to utilize a mobile application for CVD management.

Exclusion Criteria:

* A history of stroke, myocardial infarction or any related cardiovascular complications Complicated diabetes mellitus e.g., Proliferative diabetic retinopathy, end-stage renal disease
* Unavailability of a smartphone or any reason that will not allow the participant to use the app properly. (such as; difficulty or inability to use mobile applications, unavailability of network services…etc.).
* Medical conditions that restrain the participant to be physically active.
* High chance of loss to follow up at the FAMCO clinic (due to upcoming travel, temporary employment and thus eligibility to be treated at the clinic, irregular visits due to distance from home…etc.)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 410 (Estimated)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Reduced blood cholesterol and triglycerides levels | 18 months
  Immunoassay based-method will be used to measure lipid profile in the blood samples collected from the study participants. Lipids will be measured in millimole/Liter This outcome will be achieved when the Participants lipid profile is reduced compared to the initial values (measured at the beginning of the study)
  The assessment will be base don the ranges below:
  Total Cholesterol (mmol/L): < 5.2 / TG (mmol/L): (0 - 2.3) / LDL-C (mmol/L): < 2.59 / HDL-C (mmol/L): > 1.68 (Female) >1.45 (Male)
Reduced blood glucose levels | 18 months
  Glucometer devices for fasting blood glucose and for glycated hemoglobin will be used to asses the improvement in impaired glycemia.
  Participants who achieve this outcome would have reduced blood glucose compared to the initial values (measured at the beginning of the study)
  The following measures will be used to asses the glycemic state of the pateints
  Fasting blood glucose: (Norma < 5.6 mmol/L), (Impaired glycemia/type 2 diabetes ≥ 5.6 mmol/L) Glycated hemoglobin (HbA1c): (Normal < 5.7 %), (> 6.5 Diabetes)
Normalized blood pressure | 18 months
  systolic blood pressure and diastolic blood pressure of the participants will measured throughout the study using sphygmomanometer
  The measures below will be used to assess the improvement in the blood pressure of the participants Hypertension: systolic blood pressure ≥ 130 mmHg and/or diastolic blood pressure ≥ 85 mmHg Normal blood pressure: systolic: < 120 mm Hg/ diastolic < 80 mm Hg
Reduced BMI and visceral obesity | 18 months
  Anthropometric measurements (height, weight, waist and hip circumferences) will be taken from the participants throughout the study.
  Body Mass Index (BMI) will be measured using the formula BMI = weight(kg)/height(m2).
  Desired BMI is in the range of 18.5 to 24.9, A BMI of 25.0 or more is overweight
  Visceral obesity will be assed by measuring the waist-to-hip ratio Female: > 0.85 No visceral obesity, < 0.85 existing visceral obesity Male: > 1.0 No visceral obesity, < 1.0 existing visceral obesity

SECONDARY OUTCOMES:
Increased physical activity and increased intake of healthy diet | 18 months
  The daily physical activity will will be measured by pedometer feature of the mobile application in the form of number of foot steps.
  Intake of healthy diet will also be assessed using the mobile application by counting the number of vegetables/fruits servings per day.
  The overall increase in the physical activity and intake of healthy diet will be assessed during the study visits (every 4 months) using a standardized validated questionnaires namely "Dubasi questionnaire on dietary intake and physical activity". This questionnaire is based on likert score (Dubasi, S.K., et al., Questionnaire to assess adherence to diet and exercise advices for weight management in lifestyle-related diseases. J Family Med Prim Care, 2019. 8(2): p. 689-694.)
Reduced alcohol consumption and tobacco smoking | 18
  The reduction in alcohol consumption and tobacco smoking will be assessed using Standardized validated questionnaires The Fagerström test for Nicotine Dependence which asses the intensity of physical addiction to nicotine Alcohol Use Disorders Identification Test (AUDIT) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Amani Alkhaifi, PhD, Principal Investigator — Sultan Qaboos University

IPD SHARING:
Plan to Share IPD: No